CLINICAL TRIAL: NCT04322929
Title: Anti-inflammatory Effects of Roflumilast Treatment for 12 Weeks in Stable-state Non-cystic Fibrosis Bronchiectasis
Brief Title: Roflumilast in Non-CF Bronchiectasis Study (2019)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Chung-Man HO, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROF2019_v2
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Non-cystic Fibrosis Bronchiectasis
Keywords: 24-hour sputum volume; Roflumilast
MeSH Terms: interventions — Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral roflumilast (Experimental): Oral roflumilast 250 microgram daily will be started at the baseline visit for 4 weeks. For those who can tolerate the initial 4-week treatment, roflumilast will be increased to 500 microgram daily, allowing subsequent dose reduction back to 250 microgram daily in case of CTCAE grade 3 or 4 toxicities.
  Interventions: Drug: Roflumilast Oral Tablet

INTERVENTIONS:
Drug: Roflumilast Oral Tablet — Roflumilast, a phosphodiesterase 4 (PDE4) inhibitor is approved worldwide (including Hong Kong) for treatment of severe chronic obstructive pulmonary disease (COPD) with frequent exacerbations. Roflumilast has been shown to have anti-inflammatory effect in patients with COPD, with significant reduction of sputum absolute neutrophil count, IL-8 and neutrophil elastase compared with placebo treatment. Roflumilast can also improve the lung function parameters in patients with COPD and reduce the rate of moderate-to-severe exacerbations.
  Other Names: Daxas

SUMMARY:
This is a single-arm, open label, Phase II study of 12-week use of Roflumilast in stable-state non-cystic fibrosis bronchiectasis subjects.

Bronchiectasis refers to a suppurative lung condition characterized by pathological dilatation of bronchi. The predominant aetiology of bronchiectasis in the Western population is related to cystic fibrosis (CF), which is genetically determined. Bronchiectasis due to other causes are generally grouped under the term "non-CF bronchiectasis", which accounts for practically all cases that are seen commonly in Hong Kong and many other Chinese populations.

The main pathogenesis of non-CF bronchiectasis involves airway inflammation, abnormal mucus clearance and bacterial colonization, resulting in progressive airway destruction and distortion. This destructive process perpetuates in a vicious circle even when the initial insult has subsided, which is commonly due to an infective process like tuberculosis in Hong Kong. Patients with extensive bronchiectasis present with chronic cough, copious purulent sputum, haemoptysis, progressive lung function loss, and episodes of infective exacerbations.

The current treatment strategies mainly focus on targeting the key elements in the pathogenesis of non-CF bronchiectasis. Apart from regular chest physiotherapy and postural drainage to help clearing mucus from bronchiectatic airways, inhalational and parenteral antibiotics have also been used to reduce the bacterial load in destroyed airways, thus controlling and preventing infective exacerbations. In recent years, accumulated evidence has suggested a central role of airway inflammation and immune dysregulation in the evolution of non-CF bronchiectasis.

Chronic obstructive pulmonary disease (COPD) is a progressive destructive process on exposure to noxious environmental agents (e.g. tobacco smoke) that affects both the airways (chronic bronchitis) and lung parenchyma (emphysema), leading to loss of lung function and exercise capacity. Both COPD and bronchiectasis share similarities in clinical presentation and pathogenetic mechanisms. Neutrophilic inflammation and bacterial colonization are also the cornerstone in the airways of patients with COPD. Roflumilast, a phosphodiesterase 4 (PDE4) inhibitor, has demonstrated anti-inflammatory activity in COPD resulting in reduction in exacerbation frequency. This is the first-in-class and the only one clinically available PDE4 inhibitor that is approved worldwide (including Hong Kong) for treatment of severe COPD with frequent exacerbations.

At the time of writing, the exact role and clinical evidence for roflumilast in dampening airway inflammation in non-CF bronchiectasis is still lacking. Given the common pathogenetic mechanism via neutrophilic inflammation between non-CF bronchiectasis and COPD, as well as the robust clinical activity of roflumilast in COPD, this study is designed to provide initial scientific evidence on the activity of roflumilast on neutrophilic airway inflammation in patients with stable-state non-CF bronchiectasis.

This study aims to investigate the effect of 12-week treatment with roflumilast on neutrophilic airway inflammation in stable-state non-CF bronchiectasis.

DETAILED DESCRIPTION:
In a 4-week crossover study in 38 patients with COPD, roflumilast 500μg daily significantly reduced sputum absolute neutrophil count, IL-8 and neutrophil elastase compared with placebo treatment. Interestingly, the mechanism of anti-neutrophilic inflammation with roflumilast treatment in patients with COPD was recently found to be mediated through decreasing prolyl endopeptidase activity and acetyl-proline-glycine-proline (AcPGP), thus providing a clear biological plausibility for clinical activity of roflumilast. The clinical benefits of roflumilast treatment in COPD were subsequently demonstrated in 2 identical RCTs involving 3,096 patients with COPD having severe airflow limitation and history of exacerbations. Treatment with roflumilast 500μg daily resulted in better prebronchodilator FEV1 (by 48 ml in 52 weeks) and lower rate of exacerbations (reduction by 17%) compared with placebo treatment. The benefit of roflumilast on lung function has also been confirmed in another 2 identical RCTs among those patients with moderate to severe COPD already treated with long-acting bronchodilators (salmeterol or tiotropium). The mean pre-bronchodilator FEV1 was significantly improved with roflumilast compared to placebo treatment for 24 weeks by 49ml and 80ml respectively in patients with COPD already treated with salmeterol and tiotropium respectively. More recently, among patients with more severe COPD requiring combination ICS/long-acting β2 agonist, roflumilast treatment for 52 weeks significantly reduced the rate of moderate-to-severe exacerbations by 13.2% compared to placebo group. The safety and adverse effects of roflumilast have been well-tolerated, resulting in worldwide (including Hong Kong) approval for clinical use in COPD. The common adverse effects of roflumilast treatment include weight reduction (>10% loss in 7% subjects), decreased appetite (2%), insomnia (2%), headache (4%), diarrhea (10%) and nausea (5%).

Our group has previously embarked on various clinical studies in non-CF bronchiectasis: a 4-week treatment of inhaled fluticasone (ICS) compared with placebo (1), a subsequent 52-week randomized controlled trial of inhaled fluticasone in 86 patients (4), and a separate study on sputum elastase in 30 patients (2). These support the feasibility of conducting similar clinical trials, like the current proposal, on non-CF bronchiectasis in our unit. To prepare for the current study proposal, we have conducted a pilot and feasibility study of 4-week treatment of roflumilast in stable-state non-CF bronchiectasis with the exact inclusion/exclusion criteria as the current proposal (HKU/HA HKW IRB approval no. UW 17-444) since March 2018. Up to January 2019, we have successfully recruited 15 eligible study subjects. The initial study protocol mandated the starting dose of roflumilast at 500 microgram daily. The first two study subjects experienced intolerable gastrointestinal side effects within 1-2 weeks of treatment, leading to premature treatment cessation. An amended study protocol (HKU/HA HKW IRB approval dated 24 July 2018) was approved that allowed a lower initiating dose of 250 microgram daily, which is in line with the current recommended prescription in COPD patients. Nine out of the subsequent 13 subjects (including the most recent 8 subjects consecutively) were able to complete roflumilast 250 microgram daily treatment for a total of 4 weeks, with less than grade 1 toxicities. The characteristics of the nine per-protocol study subjects include: M:F=4:5, age of 69.9 ± 9.1 years (mean ± SD) and baseline 24-h sputum volume of 30.00 ± 26.93 ml (for all 15 subjects: 27.47 ± 22.59 ml). The preliminary results showed insignificant change in sputum volume and a trend of reduced sputum IL-1β (pre- vs post-treatment: 10.84 vs 2.63 ng/ml, p=0.102). This indicates a possible anti-inflammatory effect of roflumilast in non-CF bronchiectasis with just 4 weeks of treatment, though this pilot was meant for feasibility study and not powered to detect significant change. The true benefit will likely require a longer duration of treatment (thus proposing 12 weeks in this study) with sufficient sample size.

This study aims to investigate the effect of 12-week treatment with roflumilast on neutrophilic airway inflammation in stable-state non-CF bronchiectasis. The primary outcome measure is 24-h sputum volume. The extent of airway inflammation in non-CF bronchiectasis is indicated by sputum leukocyte density, pro-inflammatory cytokines (IL-1β, IL-8, TNF-alpha, LTB4 and IL-17) and neutrophil elastase. Health-related quality of life (HRQoL) is a key secondary outcome. We hypothesize that 12-week treatment of roflumilast in stable-state non-CF bronchiectasis can result in: (1) reduction in 24-h sputum volume (primary hypothesis); (2) reduction in sputum leukocyte density; (3) reduction in sputum pro-inflammatory cytokines (IL-1β, IL-8, TNF-alpha, and IL-17) and LTB4; (4) reduction in sputum neutrophil elastase; (5) no change in sputum bacterial colonization and load; (6) improvement in HRQoL.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or above, male or female.
2. Never-smokers or those who have smoked less than 100 cigarettes in their lifetime.
3. Confirmed diagnosis of non-CF bronchiectasis based on high-resolution computed tomography (HRCT) scan.
4. Significant sputum production (≥ 10 ml per day).
5. In stable-state bronchiectasis with no change in regular medications (e.g. inhaled steroid, macrolide) or exacerbations in the past 3 months.
6. Written informed consent obtained.

Exclusion Criteria:

1. Eversmokers (≥ 100 cigarettes in their lifetime).
2. Known chronic obstructive pulmonary disease or asthma.
3. Moderate to severe liver impairment (Child-Pugh B or C).
4. Known psychiatric illness with increased suicidal risks.
5. Body-mass index below 18 kg/m2.
6. Concomitant use of strong cytochrome P450 inducers (e.g. rifampicin, phenobarbital, carbamazepine, phenytoin).
7. Patients who are hypersensitive to roflumilast or its constituents.
8. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
24-hour sputum volume | Reduction in 24-h sputum volume in 12 weeks
  Daily sputum volume is determined as the average of a three consecutive day collection (9:00 a.m. to 9:00 a.m.) at home, using clear pre-labeled sterile plastic (60 ml) pots stored at 4°C. Subjects are instructed and trained to completely empty the contents of their mouth before expectorating into the sputum pots to ensure minimal contamination by saliva and food debris. The volume of a 24-hour sputum specimen is determined as the volume of water (to the nearest 0.1 ml) in an adjacent identical pot containing water at the same level as the sputum in the sputum-containing pot.

SECONDARY OUTCOMES:
Sputum leukocyte density | Reduction in sputum leukocyte density in 12 weeks
  A fresh sputum sample is collected in a sterile clear plastic pot after thorough mouth emptying on the day of planned clinic visit. Sputum leukocyte density is measured within 2 hours of collection by a designated technician, based on five aliquots chosen randomly from the center of a fresh specimen, which are then serially diluted with phosphate-buffered saline (PBS) and read with a light microscope and a hemocytometer as we previously described.
Sputum pro-inflammatory cytokines (IL-1β, IL-8, TNF-alpha, and IL-17) and LTB4 | Reduction in sputum pro-inflammatory cytokines in 12 weeks
  Fresh sputum sample is stored at -70° C within 15 min of collection until ultracentrifugation (100,000 g for 30 min at 4° C) to obtain the sol phase used for enzyme-linked immunoabsorbent assay of cytokines (IL-1β, IL-8, TNF-alpha, IL-17) and LTB4 levels using commercially available kits.
Sputum neutrophil elastase | Reduction in sputum neutrophil elastase in 12 weeks
  Sputum neutrophil elastatse is measured using a commercially available kinetic, chromogenic microtitre plate assay with succinyl-Ala-Ala-Pro-Val-p-nitroanalide (Bachem) as a substrate, as we previously described. A standard curve, constructed from known concentrations of purified elastase, is included in each assay.
Sputum bacterial colonization and load | No change in sputum bacterial colonization and load in 12 weeks
  Sputum for bacterial culture is saved and sputum bacterial load is measured at designated visits as described previously with modifications.
Health-related quality of life (HRQoL) | Improvement in HRQoL in 12 weeks
  Patients' HRQoL will be measured by St. George's Respiratory Questionnaire Hong Kong Chinese version (SGRQ-HK). SGRQ-HK is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airway disease. It consists of 2 parts with 50 items. It addresses frequency and severity patients' symptoms, as well as activities that cause or are limited by breathlessness. The scores range from 0 to 100, with higher scores indicating more limitations. The minimally important difference is a mean change of 4 units for slightly efficacious treatment, 8 units for moderately efficacious change and 12 units for very efficacious treatment. SGRQ-HK has been validated in patients with bronchiectasis and is considered a valid and sensitive instrument for determining quality of life in bronchiectasis patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No